CLINICAL TRIAL: NCT04260932
Title: CD19/CD20 Dual-CAR-T for Patients With B-cell Lymphoma
Brief Title: CD19/CD20 Dual-CAR-T in B-cell Lymphoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-006
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-08

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/CD20 Dual-CAR-T cells (Experimental): CD19/CD20 Dual-CAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of CAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 250mg/m2 for 3 days and take a rest for at least 2 days before infusion.
  Interventions: Biological: CD19/CD20 Dual-CAR-T cells

INTERVENTIONS:
Biological: CD19/CD20 Dual-CAR-T cells — CD19/CD20 Dual-CAR-T cells are prepared via lentiviral infection. 5 days prior to infusion of CAR-T cells, subjects receive fludarabine at dose 30mg/m2/day and cyclophosphamide treatment at dose 250mg/m2 for 3 days and take a rest at least for 2 days before infusion. CD19/CD20 Dual-CAR-T cells will be intravenously infused with a escalated dose of 1-6×106 cells/kg.

SUMMARY:
This is a single center, single arm, open-label, phase I study to evaluate the safety and efficacy of CD19/CD20 Dual-CAR-T cells in patients with refractory and relapsed B-cell lymphoma.

DETAILED DESCRIPTION:
This Phase I study is designed as a pilot trial evaluating the safety and efficacy of CD19/CD20 Dual-CAR-T cell therapy in subjects with refractory and relapsed B cell lymphoma. Subjects will receive cytoreductive chemotherapy with cyclophosphamide and fludarabine on days -5, -4 and -3 followed by infusion of CD19/CD20 Dual-CAR-T cells. Safety and efficacy of CD19/CD20 Dual-CAR-T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19/CD20 Dual-CAR-T cells therapy in patients with refractory and relapsed B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed and refractory B-cell lymphoma with:

   Relapsed or refractory disease after ≥2 lines of chemotherapy including rituximab and anthracycline and either having failed after autologous or allogeneic hematopoietic stem cell transplantation (ASCT);
2. Patients must have evaluable evidence of disease, including minimal residual disease (MRD);
3. Double positive expression of CD19 / CD20 in B cells;
4. Ages 1 to 80 years, including boundary values;
5. ECOG score 0-3 points;
6. Women of childbearing age (15-49 years old) must receive a pregnancy test within 7 days prior to initiation of treatment and the results are negative; male and female patients with fertility must use an effective contraceptive to ensure 3 months after discontinuation of treatment during the study period not pregnant inside;
7. Patients who voluntarily sign informed consent and are willing to comply with treatment plans.

Exclusion Criteria:

1. patients with organ failure:

   * Heart: NYHA heart function grade IV;
   * Liver: Grade C that achieves Child-Turcotte liver function grading;
   * Kidney: kidney failure and uremia;
   * Lung: symptoms of respiratory failure;
   * Brain: a person with a disability;
2. Active infections that are difficult to control;
3. Human immunodeficiency virus (HIV) positive;
4. Liver and kidney function: total bilirubin > 5 × ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 5 × ULN, serum creatinine clearance rate 60mL / min;
5. GVHD ≥ 2 or anti-GVHD treatment;
6. intracranial hypertension or unconsciousness; respiratory failure; diffuse vascular internal coagulation;
7. pregnant or lactating women;
8. The patient does not agree to use effective contraception during the treatment period and for the next 3 months;
9. Patients who participate in other clinical studies at the same time;
10. The investigator believes that there are other factors that are not suitable for inclusion or influence the subject's participation or completion of the study.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events. | 6 months
Objective remission rate(ORR) | 6 months
  The percentage of participants who achieved complete remission (CR) and partial remission over all participants.

SECONDARY OUTCOMES:
Relapse-Free Survival(RFS ) | 6 months
Overall-Survival(OS) | 6 months
Persistence of CAR-T cells in vivo | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China